CLINICAL TRIAL: NCT00798499
Title: A Multi Centre Study With no Treatment, Designed to Gain Information About the Haemophilia Patient Population
Brief Title: A Feasibility Study to Collect Data in Patients With Haemophilia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Brian Bryzinski, Senior Director Global Medical Research, Medical Science Director, AstraZeneca Pharmaceuticals - AZ US
Other Study IDs: D0960M00006
Record Dates: First submitted 2008-11-12; First posted 2008-11-26 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-07

CONDITIONS: Hemophilia
Keywords: haemophilia; patients with haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples Without DNA — plasma

GROUPS / COHORTS (1):
- 1: Laboratory variables
  Interventions: Other: Laboratory variables

INTERVENTIONS:
Other: Laboratory variables — 1 visit

SUMMARY:
The purpose of this study is to collect reference data in patients with haemophilia. The study will also collect and store blood samples for potential future exploratory research in the disease area.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients with haemophilia, all severities
* At least 18 years old.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Laboratory variables related to coagulation, SAEs in connection to blood sampling procedures will be collected, non-serious AEs will not be recorded | The variables will be measured at first visit.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Berntorp, MD, PhD, Professor, Principal Investigator — Malmo University
Locations (2):
- Sweden (2):
  - Research Site, Malmo
  - Research Site, Stockholm